CLINICAL TRIAL: NCT05930535
Title: Family-Focused Adolescent & Lifelong Health Promotion - Study Protocol of Phase 1
Brief Title: Family-Focused Adolescent & Lifelong Health Promotion
Acronym: FLOURISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Klagenfurt (Other)
Collaborators: Institute for Marriage, Family and Systemic Practice - ALTERNATIVA (Other); Health for Youth Association, Moldova (Other); Cardiff University (Other); Bielefeld University (Other); Association for Systematic Therapy Education Center (Unknown); Medical University of Vienna (Other); University Jaume I Castellon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101095528
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Behavior; Adolescent - Emotional Problem; Psychological Well-Being; Parent-Child Relations; Parenting
Keywords: Parenting; Mental health; MOST design; Adolescents; Family-based intervention
MeSH Terms: conditions — Adolescent Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All participants will be allocated to the same intervention arm for this pilot feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parenting for Lifelong Health (Experimental): Parenting Program "Parenting for Lifelong Health" (PLH) for parents and their teens aged 10-14 years old with Helping Adolescents Thrive comics at home
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens

INTERVENTIONS:
Behavioral: Parenting for Lifelong Health for Parents and Teens — PLH will be delivered over 6 sessions as a group-based family program with both adolescents and caregivers attending, with joint and separate core sessions framed by joint introductions and endings. It will include activities such as: building positive parent-child relationships; developing problem-solving skills; stress-management and stress-reduction skills; improving effective limit-setting and discipline by parents; talking about feelings and regulating emotions.
  The PLH program will also include a peer support component and incentive boosters. The Helping Adolescents Thrive comic chapters will be provided as homework activities. The comics, developed by UNICEF, cover adaptation to new situations, stress management, problem-solving, communication skills, risky choices and being there for each other.

SUMMARY:
The aim of this study is to adapt the Parenting for Lifelong Health for Parents and Teens (PLH) with the Helping Adolescents Thrive Comics in North Macedonia and the Republic of Moldova and conduct a pilot feasibility study of the adapted version. The program will be delivered by ALTERNATIVA in North Macedonia and Health for Youth Association in the Republic of Moldova.

The intervention and training materials will be adapted for the local context and languages (Romanian, Macedonian, and Russian). Facilitators and coaches will be trained to deliver the intervention in the fall of 2023. A pre-post pilot study will be conducted testing the feasibility of the program and the assessment measures with caregivers (30 per country) and their 10-14-year-old children (30 per country). This includes examination of outcomes related to implementation fidelity, program acceptability, and preliminary program effectiveness in improving teens' behavioral and emotional problems.

This feasibility study is part of a larger implementation science project using the MOST framework (Multiphase Optimization Strategy). This specific protocol is for the preparation phase of MOST (Phase 1). There are two more phases of MOST that will follow: the optimization phase (Phase 2) and the evaluation phase (Phase 3). The results of Phase 1 will be used to inform any changes to the intervention and assessment measures that may be necessary before testing the intervention in Phase 2, which will involve a randomized factorial trial.

DETAILED DESCRIPTION:
Mental health problems during early adolescence are a global concern, especially in low- and middle-income countries (LMICs). North Macedonia and the Republic of Moldova are among the poorest countries in Europe and many children in these countries are exposed to risk factors for negative mental health outcomes, such as family violence. In addition, the recent coronavirus pandemic and war in Ukraine have greatly increased economic, social, and psychological challenges in Eastern Europe. This situation makes the prevention of mental health problems and promotion of well-being among adolescents in North Macedonia and Republic of Moldova a high priority.

Parenting programs are recommended by many health guidelines as evidence-based solutions to support adolescent well-being. One example of a program developed specifically for low- and middle-income contexts is Parenting for Lifelong Health (PLH), a group-based social-behavioral intervention. However, a major challenge of implementing such programs entails sustaining and embedding them into lasting delivery systems (scaling-up). As a result, it is critical to optimize parenting programs in low-resource settings. Specifically, it is essential to identify the most effective and cost-effective components of parenting programs.

The present project, "FLOURISH", aims to adapt the Parenting for Lifelong Health for Parents and Teens (PLH) and the Helping Adolescents Thrive (HAT) Comics in North Macedonia and the Republic of Moldova and conduct a pilot feasibility study of the adapted version. The program will be delivered by ALTERNATIVA in North Macedonia and Health for Youth Association in the Republic of Moldova.

FLOURISH will consist of one clinical study with three phases (studies will be registered separately) based on the MOST framework:

Phase 1: Program adaptation and piloting (Preparation of MOST)

Phase 2: Factorial trial and process evaluation (Optimization of MOST)

Phase 3: Hybrid implementation-effectiveness randomized trial and process evaluation (Evaluation of MOST).

This protocol is for the Preparation phase of MOST and will inform the subsequent phases of the project. It consists of a pre-post evaluation testing the feasibility of the program with 30 caregivers and their children aged 10-14 years old in each country site and examining outcomes related to implementation fidelity, program acceptability, and preliminary program effectiveness in improving teens' mental health and family well-being.

The PLH for Parents and Teens program will include an adolescent peer support component and adolescent participation boosters, which are candidate components for testing in Phase 2. The peer support component will introduce a systematic strategy of social support enhancement in each intervention group. Each adolescent will pair up with another adolescent from their group.The adolescent participation boosters will involve a selection of incentives for participation that will be determined based on initial coproduction activities.

As an add-on to the PLH program and third candidate component to pilot in Phase 1, the Magnificent Mei comics as part of the Helping Adolescents Thrive materials will be provided to adolescents for at home practice. The comics consists of 6 chapters which cover the following topics: adaptation to new situations, stress management, problem-solving, communication skills, risky choices and being there for each other. We will adapt the content together with UNICEF and the advisory groups.

In addition, all study materials will be adapted into the local languages (Romanian, Macedonian, and Russian). The assessment measures will be translated following a detailed translation script. This also includes intervention cost and other health economic measures for resource use (PECUNIA RUM), health-related quality of life (EQ5D-5L, EQ5D-Y(3L)) and capability well-being (OxCAP-MH) used to evaluate costs and outcomes for the cost effectiveness analyses in Phase 2. The initial psychometric results from a mini pilot (5 adolescents and 5 caregivers for each language), as well as the pre-post outcomes during this phase, will inform decisions on measures for Phase 2.

This study will also pilot a range of measures, reported by implementation staff, to record the time and resources required for intervention delivery, document the background and well-being of frontline intervention staff, and assess the fidelity of intervention delivery, using a structured observation tool.

The pilot feasibility study will be informed by other activities during this Phase. This include coproduction advisory groups with caregivers, adolescents, intervention staff, and professional experts, context-mapping expert interviews, and post-intervention focus-groups. These activities will be informative in assessing feasibility and acceptability of the intervention and context specific adaptations.

ELIGIBILITY:
Inclusion Criteria:

1. for Caregivers:

   * Age 18 or older at baseline assessment;
   * Primary caregiver responsible for the care of an adolescent 10-14 who is a resident in the same household at least four nights a week in the previous month;
   * Able to speak at least one of the local languages in which the program will be offered (Romanian, Russian, Macedonian)
   * Agreement to participate in the program;
   * Provision of consent for self and child to participate in the study.
2. for Adolescents:

   * Age 10-14 at baseline assessment;
   * Assent to participate in the study;
   * Caregiver consent to participate in the study.

Exclusion Criteria:

No formal exclusion criteria have been set for FLOURISH. However, during the process of introducing the project, the research team will guide the participants through a consent form that asks whether they are currently experiencing acute distress or a mental health or physical health condition that would interfere with their participation. The judgement will be made by the potential participant. If the participant decides they are not currently able to take part due to acute health issues, the research team will follow up and provide referrals for other services.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Change in levels of adolescent emotional problems: Revised Child Anxiety and Depression Scales (RCADS), subscales | Pre-assessment and 6 - 8 weeks after pre-assessment
  The RCADS is a self-report measure developed to evaluate among children symptoms of a number of DSM defined anxiety and depression disorders with two subscales. The RCADS requires respondents to rate how often each item applies to them. Items are scored 0-3 corresponding to ''never,'' ''sometimes,'' ''often,'' and ''always''.
Change in levels of adolescent emotional problems: Child Behavior Checklist (CBCL) 6-18, internalizing subscale | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CBCL is an instrument from the Achenbach System of Empirically Based Assessment (ASEBA). Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of adolescent emotional problems: Youth Self-Report (YSR) 11-18, internalizing subscale | Pre-assessment and 6 - 8 weeks after pre-assessment
  The YSR is an instrument from the Achenbach System of Empirically Based Assessment (ASEBA). Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of adolescent behavior problems: Child Behavior Checklist (CBCL) 6-18, parent-report, subscales rule-breaking and aggressive behavior | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CBCL is an instrument from the Achenbach System of Empirically Based Assessment (ASEBA). The CBCL is a widely used instrument for assessing child behavioral and emotional symptoms.
  Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of adolescent behavior problems: Youth Self-Report (YSR) 11-18, child-report, subscales rule-breaking and aggressive behavior | Pre-assessment and 6 - 8 weeks after pre-assessment
  The YSR is an instrument from the Achenbach System of Empirically Based Assessment (ASEBA). These YSR is widely used for assessing child behavioral and emotional symptoms.
  Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of well-being in adolescents: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The WHO-5 is a short, positively worded instrument designed to assess the level of emotional well-being over 14 days. Respondents are asked to rate how well each of the 5 statements applies to them when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time) with a range of scores from 0 (absence of well-being) to 25 (maximum score on well-being).

SECONDARY OUTCOMES:
Change in levels of family communication in adolescents: Child-Parent Communication Apprehension scale (CPA-YA), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CPA-YA measures parent-child communication apprehension and will be completed by adolescents. The tools consists of 12 items with responses being scored using a 5-point Likert-type scale, from 1 (strongly disagree) to 5 (strongly agree).
Change in levels of family functioning in caregivers: Family Assessment Device (FAD), subscale "general functioning" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The general functioning subscale is one of the dimensions of the FAD and will be completed by caregivers. This scale has also been used as a single indicator to assess family functioning. The general functioning scale is made up of 12 items with six items that reflect healthy family functioning and the other six items reflecting unhealthy functioning. Scoring is on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scoring for the negatively worded items reversed.
Change in frequency of parenting practices: Alabama Parenting Questionnaire-APQ, subscale "involved parenting", subscale "parental supervision/monitoring " (parent- and child-report) and subscale "corporal punishment" (parent-report) | Pre-assessment and 6 - 8 weeks after pre-assessment
  Parenting practices will be assessed with the child- and parent-report version of the Alabama Parenting Questionnaire (APQ). The APQ is a self-report measure of parenting behaviors designed to assess the parenting practices most related to disruptive behaviors of children. The APQ subscales may be rated by parents and children (caregiver-report and child-report) using a 5-point scale ranging from 1 (never) to 5 (always).
Change in levels of loneliness in adolescents: UCLA-8 Loneliness scale, total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The UCLA-8 is brief 8-item version developed specifically for use with adolescents. Items are scored on 4-point scale.
Change in levels of social support in adolescents and caregivers: Medical Outcome Study Social Support Survey (MOS-SSS), "emotional and affectionate subscales" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The MOS-SSS includes 18 items with a response range from 1 (none of the time) to 5 (all of the time). The emotional and affectionate support scales comprise 11 items.
Change in levels of well-being in caregivers: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The WHO-5 is a short, positively worded instrument designed to assess the level of emotional well-being over 14 days. Respondents are asked to rate how well each of the 5 statements applies to them when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). Therefore, the raw score theoretically ranges from 0 (absence of well-being) to 25 (maximal well-being).
Change in levels of psychological distress in caregivers: Patient Health Questionnaire - 9 (PHQ-9) | Pre-assessment and 6 - 8 weeks after pre-assessment
  The PHQ-9 is a 9-item self-report questionnaire used as a continuous measure to assess depressive symptom severity. Response options on the items range from 'not at all' (0 points) to 'nearly every day' (3 points).
Change in levels of parental stress in caregivers: Parental Stress Scale (PSS), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The PSS is an 18-item self-report questionnaire. Items are rated on a 5-point Likert scale (1 = Strongly disagree, 2 = Disagree, 3 = Undecided, 4 = Agree, 5 = Strongly agree) and scores range from 18 to 90, with higher values indicating greater levels of parental stress.
Change in levels of emotional problems in adolescents: Revised Child Anxiety and Depression Scales (RCADS), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The RCADS requires respondents to rate how often each item applies to them. Items are scored 0-3 corresponding to ''never,'' ''sometimes,'' ''often,'' and ''always''.
Change in levels of adolescent behavior problems: Child Behavior Checklist (CBCL) 6-18, parent-report, subscale externalizing behavior | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CBCL is an instrument within the Achenbach System of Empirically Based Assessment (ASEBA), which are widely used assessments for child behavioral and emotional symptoms.
  Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of adolescent behavior problems: Youth Self-Report (YSR) 11-18, child-report, subscale externalizing behavior | Pre-assessment and 6 - 8 weeks after pre-assessment
  The YSR is an instrument within the Achenbach System of Empirically Based Assessment (ASEBA), which are widely used assessments for child behavioral and emotional symptoms.
  Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of loneliness in caregivers: Revised UCLA Loneliness scale (RULS-6), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The RULS-6 was developed as a short 6-item version suitable for use among adults.

OTHER OUTCOMES:
Enrollment rate | During the implementation of the intervention (Six weeks)
  will be assessed as follows:
  1. Percentage of participants who joined the study and have attended at least one group PLH session (individual enrolment for adolescents and caregivers)
  2. Percentage of families where both adolescent and caregiver attended at least one group PLH session (family enrolment).
Attendance rate | During the implementation of the intervention (Six weeks)
  will be assessed as follows:
  1. Percentage of group PLH sessions attended out of 6 (for adolescents and caregivers; individual attendance for adolescents and caregivers)
  2. Percentage of group PLH sessions attended by both adolescent and caregiver in a given family (family attendance)
  3. Percentage of catch-up PLH contact out of 6 (for adolescents and caregivers; individual catch-up contact for adolescents and caregivers)
Adolescent healthy weight: BMI; adolescent and caregiver reports | Pre-assessment and 6 - 8 weeks after pre-assessment
  Adolescent healthy weight will be assessed with caregiver and adolescents report on the adolescent's mass in kilograms and height in meters. This is not expected to change as a result of the intervention, but is assessed for sample description.
Caregiver alcohol use: The Alcohol Use Disorder Identification Test (AUDIT), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The AUDIT contains 10 questions concerning alcohol consumption, drinking behaviors, and alcohol-related problems. It is scored from 0 to 4 for each question, resulting in a total score ranging from 0 to 40.
Post-traumatic stress in caregivers: PTSD checklist for DSM-5 (PCL-5), short form, total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The 4-item version of the PCL-5 is a short form of the original PCL-5 consisting of 20 items. These are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely), with higher scores indicating greater symptom severity. The tool will be completed by caregivers.
Posttraumatic stress in adolescents: Children's Revised Impact of Event Scale (CRIES), total score and subscales | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CRIES is organized into two dimensions-intrusion (4 items) and avoidance (4 items) and a total score. The items are scored on a four-point scale: "not at all" receives 0 scores, "rarely" sums 1 point, "sometimes" adds 3 points, and "often" computes 5 points. This tool will be completed by adolescents.
Adolescent sexual risk behavior: Health Behavior in School-aged Children Study, sub-scale "sexual health" | Pre-assessment and 6 - 8 weeks after pre-assessment
  Sexual risk behavior among adolescents aged 13 and older will be assessed with a questionnaire which was developed as part of The Health Behavior in School-aged Children (HBSC) study. The questions assess the experience of sexual intercourse, the age of sexual initiation, methods used to prevent pregnancy at last intercourse and condom use at last intercourse.
Adolescent defined problems: The Top Problem Assessment | Pre-assessment and 6 - 8 weeks after pre-assessment
  The Top Problem Assessment assesses adolescents' problems they are most concerned about. They can name three problems they choose and provide numerical severity ratings on a scale ranging from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Foran, Prof., Principal Investigator — University of Klagenfurt; Yulia Shenderovich, Dr., Principal Investigator — Cardiff University; Marija Raleva, Prof., Principal Investigator — Institute for Marriage, Family and Systemic Practice - ALTERNATIVA; Galina Lesco, Prof., Principal Investigator — Cardiff University; Graham Moore, Prof., Principal Investigator — Cardiff University; Rhiannon Evans, Prof., Principal Investigator — Cardiff University; Nina Heinrichs, Prof., Principal Investigator — Bielefeld University; Judit Simon, Prof., Principal Investigator — Medical University of Vienna; Nevena Calovska, Prof., Principal Investigator — Association of Systemic Therapists Education Centre; Bojan Shimbov, Prof., Principal Investigator — University Jaume I Castellon, Spain
Locations (2):
- Health For Youth Association, Chisinau, Moldova
- Institute for Marriage, Family and Systemic Practice - ALTERNATIVA, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: Yes
The project has a detailed data management plan (DMP) that defines data sharing procedures. The DMP is provided as a deliverable to the European Commission and updated throughout the study funding period.
Supporting Information: Study Protocol
Time Frame: After completion of the study and publication of main results.
Access Criteria: Prof. Heather Foran is responsible for data management of the FLOURISH project. For information related to data sharing, please contact her at heather.foran@aau.at
URL: https://www.flourish-study.org/